CLINICAL TRIAL: NCT04417023
Title: B3 for NMD: Bench to Bedside and Back - Transformative Discoveries Leading to Improved Care in Neuromuscular Disease
Brief Title: B3 for NMD: Bench to Bedside and Back
Status: Enrolling by invitation | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: B3forNMD
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Neuromuscular Disease
MeSH Terms: conditions — Neuromuscular Diseases | interventions — L 644711

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole Blood, cerebrospinal fluid, Saliva, Skin Biopsy, and Muscle Biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: B3 for NMD: Bench to Bedside and Back — Transformative discoveries leading to improved care in Neuromuscular Disease

SUMMARY:
Background: Neuromuscular diseases (NMD) represent a broad group of rare genetic and acquired disorders, affecting over 300,000 people in Canada. Given the multiple different NMD subtypes, almost half of patients with NMD remain undiagnosed.

Objective: The purpose of this study is to identify genetic or other markers in patient biosamples (e.g. blood, muscle, skin samples), electrodiagnostic studies or imaging that may help physicians and scientists provide faster ways to diagnose patients with NMD, study disease progression, and discover underlying disease mechanisms that may lead to future NMD therapies.

Eligibility: Adults with NMD

Design: Participants will have blood and/or tissue samples, and data from clinical information, imaging, and electrodiagnostic studies collected. Sample and data collection at the Neuromuscular Center, The Ottawa Hospital may include blood, DNA, saliva, cerebrospinal fluid, urine and stool samples, skin or muscle biopsy, and routine diagnostic imaging studies such as electrodiagnostic studies, ultrasound, and magnetic resonance imaging.

DETAILED DESCRIPTION:
The B3 for NMD creates a streamlined approach to develop the Bench (preclinical and laboratory characterization) to Bedside (clinical and imaging assessment) and Back (biomarker, diagnostics and therapy development) approach to develop transformative therapies for patients with rare NMDs. This study focuses on assessing current diagnostic techniques and disease characterization of difficult-to-diagnose NMDs including Motor Neuron Disease (e.g. ALS), Neuromuscular Junction Disorders, Neuropathies, Myopathies.

Activity 1: Improve Diagnosis: Identification of rare and novel genes causing NMD with next generation sequencing and develop imaging modalities and biomarkers to aid in diagnosis.

A collaborative research team of clinicians, informaticians, and scientists has been formed to rapidly identify the genes and the autoimmune antibodies responsible for a wide spectrum of NMD present in the Canadian population, as well as to explore mechanisms causing these disorders. In addition, novel genetic and biomarker approaches are needed to facilitate diagnosis and permit the identification of mutations in novel genes, leading to discovery of the molecular mechanisms underlying the NMD disease state. Novel diagnostic techniques that examine thousands of genes (e.g. exome/genome sequencing), protein expression (e.g. RNA sequencing) and/or serum biomarkers (e.g. exosomes) will be assessed to provide a more rapid diagnosis for patients with NMD. In addition, imaging characteristics for these rare diseases (MRI, Muscle/Nerve Ultrasound/nerve conduction studies) need to be assessed and compared in order to provide an efficient, effective and cost-savings approach to diagnosis for patients with inherited or sporadic NMD.

Activity 2. Disease Characterization: Identifying pathophysiological mechanisms in NMD

Preclinical research provides the foundation for discoveries that improve lives for patients with NMD. The identification of cellular and molecular events that govern normal muscle and nerve differentiation drives the development of regenerative-based therapies, whereas the characterization of the disease state uncovers new therapeutic targets for disease intervention. Although many NMDs were previously incurable, recent breakthroughs in the molecular pathogenesis of monogenic and acquired disorders are now revealing potential targeted disease-modifying therapies that may improve muscle health and prevent disability. The goal is to assess clinical samples such as blood, skin/muscle biopsies, cerebrospinal fluid obtained through collaboration with NeuroMuscular Centre clinicians and researchers to help develop effective novel/known drug compounds that may act as promising therapies that, in the future, can be rapidly moved into local and multicenter clinical trials.

ELIGIBILITY:
Inclusion Criteria:

Patients or blood relatives of patients classified as having a neuromuscular disease from the following categories:

* Motor Neuron Disease (Amyotrophic Lateral Sclerosis/Spinal Muscular Atrophy)
* Neuropathies
* Neuromuscular Junction Disorders
* Myopathies.

Exclusion Criteria:

Patients referred to the neurology clinic without a neuromuscular disorder:

* Central nervous system disorders such as Stroke
* Multiple Sclerosis
* Parkinson's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Affected or unaffected cohorts (including genetic carriers or non-carriers as reference biospecimens
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
To provide a more rapid diagnosis for patients with rare NMD and identify NMD biomarkers. | 5 years
  Identification of genes responsible for rare genetic NMD diseases, biomarkers, and imaging techniques to aid in diagnosis and disease management.
  Genetic and Biomarker Samples: 5 to 10 ml of blood or saliva will be collected preferably during routine medical care for DNA extraction. Urine or other bodily fluid collection will be used for biomarker studies. Fibroblast or myoblast samples can be used to establish a cell line. Unaffected family members can also provide tissue samples for DNA extraction or establishment of cell lines that will be stored in the Ottawa Hospital Neuromuscular Biobank.
  Imaging: Routine diagnostic imaging studies will be analyzed for pattern of involvement: Electrodiagnostic Studies (Nerve Conduction and Electromyogram Studies) will be included to assess nerve and muscle dysfunction, Ultrasound images of affected muscles and nerves, and MRI whole-body scans will be obtained for whole muscle qualitative evaluation and to assess inflammation and edema

SECONDARY OUTCOMES:
To characterize disease mechanisms to advance potential therapies of tomorrow. | 5 years
  Disease Characterization: Functional validation of gene candidates
  Genetic Diagnosis: Disease-causing genetic variants must be proven with genetic or functional data. Biochemical validation of a putative pathological variant to confirm the functional significance of a newly identified mutation can be considered confirmatory in some cases.
  Biomarker Development: We will use patient-derived material to develop biomarkers using metabolomic, proteomic, and transcriptional profiling. We will perform computational and in vitro screens using system-wide RNA and chemical libraries to look for modifications of disease-specific biomarkers.
  Sample analysis: We developed a collaborative network of laboratory-based scientists at the Ottawa Hospital Research Institute, University of Ottawa Faculty of Medicine, and the Children's Hospital of Eastern Ontario, and across Canada. This is vital to the validation of gene candidates and biomechanical mechanisms for the diagnosis or rare dis

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jodi Warman Chardon, MD PhD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No